CLINICAL TRIAL: NCT04111445
Title: First-in-human (FIH), Open-Label, Phase I (Dose Escalation) Study of ADG116 in Patients With Advanced/Metastatic Solid Tumors
Brief Title: Study of ADG116 in Patients With Advanced/Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study discontinued due to business decision.
Sponsor: Adagene Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG116-1001
Record Dates: First submitted 2019-09-11; First posted 2019-10-01 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADG116 (Experimental)
  Interventions: Drug: ADG116

INTERVENTIONS:
Drug: ADG116 — IV infusion at Day 1 of each cycle

SUMMARY:
This is a FIH, open-label, Phase I dose-escalation study of ADG116 in subjects with advanced/metastatic solid tumors. Study drug, ADG116, is an anti -CTLA-4 fully human monoclonal antibody that specifically binds to human CTLA-4. ADG 116 administered intravenously (IV) over a period of 60-90 minutes. The study planned to treated 42 patients.

ELIGIBILITY:
Inclusion Criteria

* Male or female, 18-75 years of age at the time of consent.
* Provide written informed consent.
* Subjects with advanced and/or metastatic histologically or cytologically confirmed solid tumor who have not responded or progressed after standard therapies or for whom no further standard therapy exists or standard therapy is not available
* Patients who are refractory or relapsed to prior anti-CTLA4 checkpoint inhibitors will also be recruited if they meet all eligibility criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* Adequate organ and bone marrow function
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within the 7 days prior to study

Exclusion Criteria:

* Pregnant or nursing females.
* Treatment with any investigational drug within 4 weeks prior to the first dose of study drug
* Grade ≥ 3 immune-related adverse events (irAE) or irAE that lead to discontinuation of prior immunotherapy. Untreated or uncontrolled central nervous system (CNS) tumors or metastases
* Any active autoimmune disease or documented history of autoimmune disease.
* Infection of human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Subjects requiring systemic treatment with corticosteroids or other immunosuppressive medications within 21 days before the planned first dose of study drug.
* Current or prior history of pneumonitis, hepatitis, nephritis, colitis or thyroiditis. Peripheral neuropathy ≥ Grade 2.
* History of clinically significant cardiac disease.
* Uncontrolled current illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities | From first dose of ADG116 (Week 1 Day 1) until 30days after the last ADG116 injection (up to 2 years)
Number of participants experiencing clinical and laboratory adverse events (AEs) | From first dose of ADG116 (Week 1 Day 1) until 30days after the last ADG116 injection (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- NEXT Oncology, San Antonio, Texas, United States